CLINICAL TRIAL: NCT03497611
Title: Edwards SAPIEN 3 PPI Registry - A Retrospective Survey and Prospective Identification of Procedure Related Variables Associated With Permanent Pacemaker Implantation in Patients Receiving an Edwards SAPIEN 3 Valve
Brief Title: Edwards SAPIEN 3 PPI Registry
Acronym: Conduct
Status: Completed | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: Conduct
Record Dates: First submitted 2018-03-26; First posted 2018-04-13 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Aortic Valve Stenosis; AV Block; Bundle-Branch Block
Keywords: Transcatheter aortic valve implantation; Pacemaker; Aortic valve calcification; PPI
MeSH Terms: conditions — Aortic Valve Stenosis; Atrioventricular Block; Bundle-Branch Block; Aortic Valve, Calcification of | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with aortic stenosis: Patients receiving Edwards SAPIEN 3 Transcatheter aortic valve implantation
  Interventions: Procedure: transcatheter valve implantation

INTERVENTIONS:
Procedure: transcatheter valve implantation — aortic transcatheter valve implantation using Edwards SAPIEN 3 valve

SUMMARY:
There are patient related risk factors for PPI that can be identified and assessed in retrospective pooling of 1000+ TAVI patient datasets.

Retrospective pooling of 6 datasets already available at participating centres (4 sites in Germany, 1 in Zwolle / The Netherlands, 1 in Linköping / Sweden).

Additional assessment of calcifications using a CT data core lab. Statistical analysis of the obtained dataset with respect to the objectives of the registry.

DETAILED DESCRIPTION:
Permanent pacemaker implantation is a widely recognized clinical event associated with TAVI becoming evident within a few days after the procedure.

While a number of registries have documented the rates of PPI with different valves, much less evidence has been provided for 1) patient based characteristics (e.g. RBBB etc.) affecting the likelihood of PPI and for 2) procedural variables (e.g. implantation depth, valve size etc.) that should be considered to perform an as safe and minimal invasive procedure as possible.

Prior research To date there are 7 published reports on pacemaker rates and predictors associated with the use of the Edwards SAPIEN 3 THV (see Table). These studies suggest that the need for pacemaker implantation in single centers ranges between 14.4 and 20.4% derived from patient numbers between 131 and 335. These analyses resulted in the identification of pre-existing conduction disturbance / aortic valve calcification as patient related and implantation depth /oversizing as procedure related variables associated with Edwards SAPIEN 3 THV TAVI. Furthermore a scoring algorithm for patient related factors has been proposed from a dataset of 240 patients to predict the likelihood of PPI after THV .

Limitations of prior research Current evidence though is limited by patient numbers versus event rates (with a max. of 62 PPI considered in any of the available datasets) resulting in a limited power in multivariable analyses, the single center design of these ventures, the lack of a consistent definition of variables potentially associated and the unexplained differences in the number and type of variables identified.

Aims For this reason the investigators consider it necessary to 1) to retrospectively pool data from all of these 7 datasets to arrive at a more comprehensive picture of patient related variables (retrospective part I), to 2) assess procedural variables in a prospective multicenter registry (prospective part II) and 3) to potentially validate the identified variables in a future prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients that already underwent Edwards SAPIEN 3 implantation because of aortic stenosis

Exclusion Criteria:

* Patients with prior pacemaker or intended valve in valve implantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that already underwent transfemoral transcatheter valve implantation with the SAPIEN 3 valve
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2018-11-03 (Actual); Study Completion 2019-03-03 (Actual)

PRIMARY OUTCOMES:
occurence of PPI after TAVI | 30 days
  need for permanent pacemaker implantation after TAVI

SECONDARY OUTCOMES:
Timing of PPI | 30 days
  Time interval after TAVI until PPI in days
Indications for PPI | 30 days
  possible reasons to implant a PP:
  * 1° AV block
  * complete RBBB
  * complete LBBB
  * QRS duration prolonged
  * LVOT calcium volume below the left and right cusp
  * etc

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Geisler, Prof., Principal Investigator — University Clinic Tübingen, Tübingen, Germany - Department of Internal Medicine III
Locations (4):
- Germany (4):
  - University Clinic Tübingen, Department of Internal Medicine III, Tübingen, Baden-Wurttemberg
  - University Clinic Ulm, Department of Internal Medicine II, Ulm, Baden-Wurttemberg
  - Herzzentrum, Universität Köln, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Münster, Klinik und Poliklinik für Erwachsene mit angeborenen und erworbenen Herzfehlern, Münster, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No
no IPD will be made available

REFERENCES:
- [Result] Droppa M, Rudolph TK, Baan J, Nielsen NE, Baumgartner H, Vendrik J, Froehlich M, Borst O, Wohrle J, Gawaz M, Potratz P, Hack LP, Mauri V, Baranowski J, Bramlage P, Kurucova J, Thoenes M, Rottbauer W, Geisler T. Risk factors for permanent pacemaker implantation in patients receiving a balloon-expandable transcatheter aortic valve prosthesis. Heart Vessels. 2020 Dec;35(12):1735-1745. doi: 10.1007/s00380-020-01653-6. Epub 2020 Jun 26. PMID 32591894
- [Derived] Rudolph T, Droppa M, Baan J, Nielsen NE, Baranowski J, Hachaturyan V, Kurucova J, Hack L, Bramlage P, Geisler T. Modifiable risk factors for permanent pacemaker after transcatheter aortic valve implantation: CONDUCT registry. Open Heart. 2023 Feb;10(1):e002191. doi: 10.1136/openhrt-2022-002191. PMID 36750275